CLINICAL TRIAL: NCT06933576
Title: Contribution of the EyeMAX™ 11Fr (Micro-Tech) Digital Single-Operator Cholangioscope With a Wide Working Channel: A Multicenter Pilot Study on the First French Experiences.
Brief Title: Contribution of the EyeMAX™ 11Fr (Micro-Tech) Digital Single-Operator Cholangioscope With a Wide Working Channel
Acronym: EyeMAX-CREGG
Status: Completed | Type: Observational
Sponsor: Clinique Paris-Bercy (Other)
Responsible Party: Principal Investigator, DAVID KARSENTI, Study coordinator, Clinique Paris-Bercy
Other Study IDs: EyeMAX-CREGG
Record Dates: First submitted 2025-04-10; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Cholangiocarcinoma; Biliary Stenosis; Bile Duct Stones; Bile Duct Stenosis
Keywords: cholangioscopy; Digital Single-Operator Cholangioscope
MeSH Terms: conditions — Cholangiocarcinoma; Cholecystolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients scheduled for cholangioscopy: All patients who underwent digital single-operator cholangioscopy using the new EyeMAX™ 11Fr (Micro-Tech Endoscopy, Nanjing, China) and were admitted to one of the CREGG centers between February 2024 and January 2025.
  Interventions: Device: DSOC EyeMAX 11Fr

INTERVENTIONS:
Device: DSOC EyeMAX 11Fr — digital single-operator cholangioscopy using the new EyeMAX™ 11Fr (Micro-Tech Endoscopy, Nanjing, China)

SUMMARY:
Background and aims Digital single-operator cholangioscopy (DSOC) enhances biliary stricture diagnosis, but the collection of quality samples can be difficult due to the small diameter of the working channel. A new DSOC (EyeMAXTM 11Fr, Micro-Tech Endoscopy, Nanjing, China) with a 2.0 mm working channel, accommodating pediatric forceps (1.6 mm), has been introduced in France. This study reports on the initial French experience.

Methods A retrospective multicenter observational study on DSOC was conducted across five endoscopy units within the CREGG (French Society of Private Hepato-Gastroenterology). Satisfaction and procedural evaluations were recorded using a visual analog scale (VAS) and compared with the SpyglassTM DS II DSOC (Boston Scientific).

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients who were referred to one of the participating expert tertiary endoscopy units for an ERCP for a bile duct stenosis

Exclusion Criteria:

* patients with significant tissue mass that could easily be punctured by EUS-FNB were not included.
* non-accessibility to the bile duct due to a history of Billroth II or Roux-en-Y reconstruction,
* coagulation disorders (such as partial thromboplastin time > 42 seconds, prothrombin time [Quick value] < 50%, or platelet count < 50,000/mm³), or treatment with clopidogrel.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study included all consecutive patients who were referred to one of the participating expert tertiary endoscopy units (5 centers from the CREGG - French Society of Private Hepato-Gastroenterology, in which the EyeMAX DSOC systems were made available), during the first year of availability of this device in France
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
overall satisfaction with the EyeMAX 11Fr DSOC | At the end of the procedure
  evaluated using a VAS (ranging from 0 - not at all satisfied - to 10 - extremely satisfied)
overall satisfaction with the EyeMAX 11Fr DSOC | At the end of the procedure
  Satisfaction with the EyeMAX 11Fr DSOC compared with the device currently available in France, the SpyGlass™ DS II DSOC. Satisfaction was categorized as better, equivalent, or worse relative to the SpyGlass™ DS II.

SECONDARY OUTCOMES:
Satisfaction of introduction of the EyeMAX 11Fr into the duodenoscope's working channel | At the end of the procedure
  Step of the procedure evaluated using a VAS (ranging from 0 - impossible - to 10 - extremely easy)
Satisfaction of the exit of the device from the working channel | At the end of the procedure
  Step of the procedure evaluated using a VAS (ranging from 0 - impossible - to 10 - extremely easy)
Satisfaction of the biliary cannulation through the papilla | At the end of the procedure
  Step of the procedure evaluated using a VAS (ranging from 0 - impossible - to 10 - extremely easy)
Satisfaction of the progression through the bile duct | At the end of the procedure
  Step of the procedure evaluated using a VAS (ranging from 0 - impossible - to 10 - extremely easy)
Satisfaction of the maneuverability | At the end of the procedure
  Step of the procedure evaluated using a VAS (ranging from 0 - impossible - to 10 - extremely easy)
Satisfaction of the ease of introducing the biopsy forceps to the target | At the end of the procedure
  Step of the procedure evaluated using a VAS (ranging from 0 - impossible - to 10 - extremely easy)
Satisfaction of the ease of performing biopsies | At the end of the procedure
  Step of the procedure evaluated using a VAS (ranging from 0 - impossible - to 10 - extremely easy)
image quality (definition, lens cleaning quality, and brightness) | At the end of the procedure
  assessed using a VAS (ranging from 0 - very poor - to 10 - exceptional)
Utility of use of the harness model compared with the model fixed directly on the duodenoscope | At the end of the procedure
  evaluated by the question: "Does the harness facilitate handling? (Y/N)"
total ERCP duration | At the end of the procedure
  described in minutes
Total cholangioscopy duration | At the end of the procedure
  described in minutes
Cholangioscopy success rate | At the end of the procedure
  Percentage of patients in whom the procedure was performed with effective bile duct visualization
Number of biopsies performed | At the end of the procedure
  Number of bile duct biopsies performed during DSOC procedure
Time required to perform biliary biopsies using DSOC | At the end of the procedure
  Described in minutes
Malignant or benign status of the biliary stricture | After more than 6 months of follow-up in cases where specimens were negative for malignancy
  The diagnosis of cholangiocarcinoma was established through biliary cytopathological examination of biopsies obtained during DSOC , biliary brushing, EUS-FNB, or surgical resection, and/or based on tumor progression observed after more than 6 months of follow-up in cases where specimens were negative for malignancy

OTHER OUTCOMES:
Adverse effects (AEs) and severe AEs due to ERCP | Within one month of the procedure
  Defined and graded according to the AGREE classification

CONTACTS AND LOCATIONS:
Overall Officials: David Karsenti, MD, Study Chair — Pôle Digestif Paris-Bercy, Clinique Paris-Bercy
Locations (5):
- France (5):
  - Clinique Paris-Bercy, Charenton-le-Pont
  - Louis Pasteur Clinic, Essey-lès-Nancy
  - Jean Mermoz Private Hospital, Lyon
  - Jules Verne Clinic, Nantes
  - Arnaud Tzang Institut, Saint-Laurent-du-Var

IPD SHARING:
Plan to Share IPD: Undecided
At this time, no decision has been made regarding the sharing of individual participant data (IPD).
  This study is the first French experience with the EyeMAX™ 11Fr digital single-operator cholangioscope and has been designed as an observational study. Accordingly, IPD sharing is not currently planned as part of the initial protocol, but may be considered at a later stage.

REFERENCES:
- [Derived] Karsenti D, Sportes A, Leblanc S, Bechet S, Derman J, Fassler I, Brieau B. Contribution of the EyeMAX 11Fr (Micro-Tech) digital single-operator cholangioscope with a wide working channel: a multicenter pilot study on the first French experiences. Therap Adv Gastroenterol. 2025 Aug 12;18:17562848251360117. doi: 10.1177/17562848251360117. eCollection 2025. PMID 40808865